CLINICAL TRIAL: NCT05058716
Title: Our Study Will be Carried Out in Hacettepe University Anesthesiology and Reanimation Intensive Care Unit. COVID-19 Positive or Suspected Patients Will be Admitted to the Unit. Coenzyme Q10 Levels Will be Checked in the First Day of Hospitalization and Once a Week. The Relationship Between Results and Clinical Course Will be Evaluated.
Brief Title: Assessment of Clinical Effects of Coenzyme Q10 Levels in COVID-19 Patients in Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Merve Goknur Soysal Kaya, Research assistant, Hacettepe University
Other Study IDs: 19423
Record Dates: First submitted 2021-09-22; First posted 2021-09-28 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 positive patients
  Interventions: Diagnostic Test: blood sample
- COVID-19 negative patients
  Interventions: Diagnostic Test: blood sample

INTERVENTIONS:
Diagnostic Test: blood sample — weekly blood sample - coenzym q10 levels

SUMMARY:
The study will be done in Hacettepe University Anesthesiology and Reanimation Intensive Care Unit. The investigators will accept COVID-19 diagnosed or suspected patients to the ICU. In the first day of hospitalization and after that once a week, the investigators will take blood samples from the patients to evaluate Coenzyme q10 levels. Our hypothesis is that there is a relationship between low coenzyme q10 levels and poor clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* being under the age of 18
* being pregnant
* patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hacettepe University Anesthesiology and Reanimation Intensive Care Unit
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
mortality | from the first day of hospitalization until the date of death from any cause
  yes or no
duration of mechanical ventilation | from the first day of hospitalization and during ICU stay period
  days
duration of vasopressor agent requirement | from the first day of hospitalization and during ICU stay period
  days

SECONDARY OUTCOMES:
any organ failure | from the first day of hospitalization until the date of death from any cause or discharge from ICU
  yes or no
new thromboembolic event | from the first day of hospitalization until the date of death from any cause or discharge from ICU
  yes or no
ICU stay period | from the first day of hospitalization until the date of death from any cause or discharge from ICU
  days
hospital stay period | from the first day of discharge from ICU to ward until the date of death or discharge from the hospital
  days

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Hospital, Ankara, Altındağ, Turkey (Türkiye)